CLINICAL TRIAL: NCT00202059
Title: The Effects of Zoledronic Acid (Zometa) and Physical Activity on Bone Density in Women Receiving Chemotherapy for Breast Cancer
Brief Title: Effects of Zometa and Physical Activity on Bone Density in Women Receiving Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1769-03-A; CZOL446E
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Bone mineral density; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid
Behavioral: Physical activity intervention

SUMMARY:
The purpose of this study is to evaluate the effect of zoledronic acid and physical activity on preventing bone loss in women aged 40 - 55 who are receiving chemotherapy for breast cancer. The primary objective is to compare the percent change in the lumbar spine bone mineral density (BMD) from baseline to 12 months for women who are randomized to either: Group A) intravenous zoledronic acid, oral calcium carbonate, and vitamin D, or Group B) a prescribed physical activity program, oral calcium carbonate and vitamin D.

DETAILED DESCRIPTION:
Background: Breast cancer diagnosis accounts for 32% of all new cancer cases in US women, with approximately 211,300 women diagnosed in 2003. The majority of these women receive adjuvant chemotherapy, which may lead to chemotherapy-induced menopause (CIM) in premenopausal women. CIM often leads to accelerated bone loss, osteopenia, and eventual osteoporosis.

Purpose: The purpose of this study is to evaluate the effect of zoledronic acid and physical activity on preventing bone loss in women aged 40 - 55 who are receiving chemotherapy for breast cancer. The primary objective is to compare the percent change in the lumbar spine bone mineral density (BMD) from baseline to 12 months for women who are randomized to either: Group A) intravenous zoledronic acid, oral calcium carbonate, and vitamin D, or Group B) a prescribed physical activity program, oral calcium carbonate and vitamin D. Secondary objectives are to compare the percent change between the groups in total hip BMD, the incidence of vertebral fractures, fatigue, functional status, and other cancer-related symptoms between the two groups.

Methods: Seventy-two women will be enrolled and randomized to one of two treatment groups. For participants randomized to Group A, intravenous zoledronic acid will be given every 3 months for the 12 month study period, along with 2 tablets of calcium carbonate (600 mg)/vitamin D (200 IU) daily. For participants randomized to Group B, a physical activity intervention designed to improve BMD will be prescribed and administered through the occupational rehabilitation department. Group B participants will also take 2 tablets of calcium carbonate (600 mg)/vitamin D (200 IU) daily. BMD measurements at the lumbar spine and hip, and an AP and lateral X-ray will be done at baseline and at 12 months after enrollment in the study, using dual energy X-ray absorptiometry (DXA). Serum bone-specific alkaline phosphotase, and N-telopeptide urine tests will be conducted at baseline and 12 months to evaluate bone resorption activity. Other measures that will be assessed via questionnaires include fatigue (Schwartz Cancer Fatigue Scale), functional status (SF-36), a 4-day food record, and other cancer-related symptoms (MD Anderson Symptom Inventory).

Analysis: Results will be analyzed on an intent-to-treat basis. Descriptive statistics will be used to analyze demographic data, tumor information, dietary information and baseline BMD. Differences between baseline means will be analyzed by t-tests. The percent change in BMD between the two groups will be analyzed by analysis of covariance (ANCOVA). Differences in other measures will be analyzed by t-tests.

Results: Results of this study will be used to determine if zoledronic acid or physical activity affect BMD in young women who are receiving chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with Stage I - II breast cancer
* Ages 40 - 55
* Pre- or peri-menopausal
* Within 1 month of beginning adjuvant or neoadjuvant chemotherapy
* Baseline lumbar spine and total hip BMD > -2.0 SD
* Able to read and write English
* Signed consent form

Exclusion Criteria:

* Previous treatment with bisphosphonates
* Laboratory evidence of renal disease
* Previous TRAM flap reconstructive surgery
* Positive pregnancy test
* Mental illness that precludes the patient from giving informed consent
* Laboratory evidence of hepatic disease

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density from baseline to 12 months after beginning chemotherapy

SECONDARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Swenson, RN, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Institute, Saint Louis Park, Minnesota, United States

REFERENCES:
- [Result] Swenson KK, Nissen MJ, Anderson E, Shapiro A, Schousboe J, Leach J. Effects of exercise vs bisphosphonates on bone mineral density in breast cancer patients receiving chemotherapy. J Support Oncol. 2009 May-Jun;7(3):101-7. PMID 19507458
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716